CLINICAL TRIAL: NCT03014076
Title: Phase Ib Trial of Combination Immunotherapy With HER2/Neu Peptide GP2 + GM-CSF Vaccine and Trastuzumab in Breast Cancer Patients
Brief Title: Immunotherapy Vaccine and Herceptin in Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cancer Insight, LLC (Industry)
Responsible Party: Principal Investigator, George E. Peoples, CEO/Founder, Cancer Insight, LLC
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C.2008.146
Record Dates: First submitted 2017-01-04; First posted 2017-01-09 (Estimated); Last update posted 2017-01-09 (Estimated); Status verified 2017-01

CONDITIONS: Breastcancer
MeSH Terms: interventions — Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GP2 peptide + GM-CSF + trastuzumab (Experimental): HLA-A2+/A3+ subjects receive GP2 + GM-CSF vaccine and trastzumab
  Interventions: Drug: GP2 peptide + GM-CSF vaccine plus trastuzumab
- Trastuzumab (Active Comparator): HLA-A2-/A3- subjects followed as controls receiving trastuzumab.
  Interventions: Drug: Trastuzumab

INTERVENTIONS:
Drug: GP2 peptide + GM-CSF vaccine plus trastuzumab — HLA-A2+/A3+ subjects are given the GP2 peptide vaccine plus trastuzumab
  Arms: GP2 peptide + GM-CSF + trastuzumab
Drug: Trastuzumab — HLA-A2-/A3- patients are followed as controls receiving trastuzumab only.
  Other Names: Herceptin
  Arms: Trastuzumab

SUMMARY:
The purpose of this trial is to determine if combination immunotherapy with HER2/neu GP2 peptide + GM-CSF vaccine and trastuzumab is safe and immunologically effective in treatment of patients with HER2/neu over-expressing breast cancer in the adjuvant setting. While not a primary endpoint, time to recurrence is measured for enrolled subjects. The objectives of the study are the following:

* Assess safety and document local and systemic toxicity to combination immunotherapy with GP2 peptide + GM-CSF vaccine and trastuzumab
* Evaluate the in vitro and in vivo immunologic responses to combination immunotherapy of GP2 peptide + GM-CSF vaccine and trastuzumab
* Determine maximum tolerated dose and optimal biologic dose for the combination immunotherapy of GP2 peptide + GM-CSF vaccine and trastuzumab

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* HER2/neu+ over-expressing breast cancer (IHC 3+ or FISH ≥2.0)
* Patients who are receiving adjuvant trastuzumab as standard of care treatment
* Completion of breast cancer therapy (i.e., surgery, radiation, and chemotherapy as appropriate per standard of care for patients' specific cancer) to exclude trastuzumab (Patients on oral hormonal therapy as part of their adjuvant breast cancer treatment will be maintained on their regimens.)
* Enrollment must occur so that patients' trastuzumab treatment and vaccine schedule overlap for all 6 vaccinations and so that first vaccination occurs after a standard of care Multiple Gated Acquisition Scan (MUGA)
* ECOG performance status (PS) 0-1
* Clinically cancer-free (no evidence of disease; excluding +CTC)
* If the patient is of childbearing potential, she must be willing to practice adequate contraception through the study treatment period and for 2 months after completion of the injection sites
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Clinical and/or radiographic evidence of residual or persistent breast cancer
* Receiving immunosuppressive therapy to include methotrexate or steroids (note: the use of prednisone, or equivalent, <2.0mg/day, is allowed)
* Tbili >1.8, creatinin >2, hemoglobin <10, platelets <100,000/mm³, WBC <2,000
* Active pulmonary disease requiring medication to include multiple inhalers
* Patients may not be receiving any other investigational agents (except with permission of the Lead Principal Investigator)
* Pregnant or are nursing
* History of autoimmune disease (patients with vitiligo not excluded)
* HIV positive
* Previous or concomitant malignancies at other sites, except effectively treated non- melanoma skin cancers or carcinoma in situ of the cervix or effectively treated malignancy that has been in remission for over 5 years and highly likely to have been cured
* Other concurrent severe medical problems, unrelated to the malignancy, that would significantly limit full compliance with the study or expose the patient to unacceptable risk
* Uncontrolled congestive heart failure or hypertension, unstable heart disease (coronary artery disease or myocardial infarction) or uncontrolled arrhythmia at the time of enrollment
* Psychiatric, addictive, or any disorder which compromises ability to give truly informed consent for participation in this study or adequate compliance

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-01; Primary Completion 2016-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Treatment-Related Adverse Events as Assessed by CTCAE v4.0 | 12 months
  Patients receiving treatment will be followed from baseline to completion of study for adverse events using CTCAE v4.0

CONTACTS AND LOCATIONS:
Overall Officials: George E Peoples, MD, Principal Investigator — Cancer Insight

IPD SHARING:
Plan to Share IPD: No